CLINICAL TRIAL: NCT03657888
Title: The Effectivenes of Family Club Denmark #Strongertogether
Acronym: FCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VIVE - The Danish Center for Social Science Research (Other)
Collaborators: KFUMs Sociale Arbejde (Unknown); FDF (Unknown); KFUM spejderne (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: VIVE100726
Record Dates: First submitted 2018-08-29; First posted 2018-09-05 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Vulnerable Families
Keywords: Family; Vulnerable; Volunteer; Child; Civil society; Intervention

STUDY DESIGN:
Intervention Model Description: The study is a prospective controlled trial with two conditions: (1) intervention group participating in Family Club Denmark and (2) wait-list control group.
Who Masked: Outcomes Assessor
Masking Description: Participants and volunteers cannot be blinded but data analyst will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family Club Denmark (FCD) (Experimental): Participation in FCD
  Interventions: Behavioral: Family Club Denmark (FCD)
- Wait-list (Other): Wait-list control
  Interventions: Other: Wait-list control

INTERVENTIONS:
Behavioral: Family Club Denmark (FCD) — Participation in Family Club Denmark
  Arms: Family Club Denmark (FCD)
Other: Wait-list control — Participants on the waiting list
  Arms: Wait-list

SUMMARY:
The aim of the trial is to assess the effectiveness of the volunteer intervention Family Club Denmark (FCD)

DETAILED DESCRIPTION:
The aim of the trial is to assess the effectiveness of the volunteer intervention Family Club Denmark (FCD). Participants are 200 vulnerable families with children aged 2-12 years, who would like to participate in a family club.

The study is a prospective controlled trial with two conditions: (1) intervention group participating in Family Club Denmark and (2) wait-list control group. Participants are allocated to intervention after a first-come-first-serve principle. When the maximum number of participants in a specific family club is reached, any further families will join the wait-list and be offered participation after 6 months.

Most participating families will be characterized by at least one of the following:

* Single parent
* Small or no network
* Low level of support
* Low income
* Physical or mental health problem
* Unemployed
* Loneliness
* Lack of contact with other adults
* Difficulty with creating relationships
* Having a hard time making ends meet during the week

A family club consists of up to 9 families. Most families are vulnerable but each club also includes nun-vulnerable families. The club is run by 3-6 volunteers who have received a 1-day training. Participants meet every two weeks for 6 months (12 sessions).

FCD is based on four principles: 1. Meal community; 2. Play, learning, and togetherness; 3. Support and advice; 4. Bridging to the civil society and the public sector

The 12 sessions center around 7 value posters:

1. Fun with smiles
2. Together but not in line
3. The time is now
4. Notice and say thank you
5. More than me
6. Courage to dare
7. Taste the world Data are collected at baseline, and after 6 and 12 months. The study is conducted in the Region South in Denmark.

ELIGIBILITY:
Inclusion Criteria:

* Family with at least one child 2-12 years old.

Exclusion Criteria:

* Not able to fill out questionnaires in Danish

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 509 (Actual)
Dates: Start 2018-09-13 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Warwick-Edinburgh Mental Well-being Scale (WEMWBS) | 6 months
  WEMWBS is a 7 item measure of maternal mental health. A total score is calculated by summing the 7 items and converting the raw score according to a published conversion table. Score range 7- 35 for both raw and converted scores. High score is better outcome.

SECONDARY OUTCOMES:
Parent Behavior Inventory (PBI) | Baseline, 6 and 12 months
  (PBI) is a 20 item that measure parenting behaviors in parents of early school-aged children. The PBI includes two subscales with high internal consistency: supportive/engaged (α =.83) and hostile/coercive (α =.81). The PBI has adequate test-retest reliability (r = .69-.74) in an ethnically diverse sample of mothers. To reduce the total number of items we include 10 items - 5 from each of the two subscales: Supportive/Engaged: items 6, 10, 11, 12, 14, and Hostile/Coercive: items 5, 9, 15, 17, 20. Score range is 0-25 for each subscale. High score is better for Supportive/Engaged, low score is better for Hostile/Coercive.
Parental Stress Scale (PSS) | Baseline, 6 and 12 months
  PSS is an 18 item measure of parenting stress that is rated on a five-point scale (Strongly disagree, Disagree, Undecided, Agree, Strongly agree). We use the revised Danish version with 16 items where the original items 2 and 11 are left out. The Danish version consists of two subscales: Parental Stress (9 items) and Lack of Parental Satisfaction (7 items). Responses are reversed for the lack of parental satisfaction items, and all responses for all items are dichotomized (0-1) before scoring. Total score range 0-9 (Parental Stress subscale) and 0-7 (Lack of Parental Stress subscale). A low score is better for both subscales.
General self-efficacy scale (GSE) | Baseline, 6 and 12 months
  GSE is a 10 item measure of optimistic self-beliefs to cope with a variety of difficult demands in life. To reduce the total number of items we include 3 items (8,9, and 10). Score range is 3-12, high score is better.
Self-worth | Baseline, 6 and 12 months
  We use 3 items from the HBSC project to measure self-worth. The 3 items are inspired by Rosenbergs concept of self-esteem. Items are scored from 1 (completely disagree) to 5 (completely agree) and summed. High score is better.
Family routines | BAseline, 6 and 12 months
  We use 5 items (1,4,9,11,21) from the Child Routine Inventory (CDI - 39 item version). Item 1,3,4, and 5 are from the Daily Living Routines subscale and item 2 is from the Household Responsibilities subscale. Inspired by the CDI we developed 5 extra items on family routines around mealtimes and language. Items are scored from 0 (never) to 4 (always). High score is better.
Kidscreen-10 | Baseline, 6 and 12 months
  Kidscreen-10 is a 10 item measure of child well-being (health-related quality of health). Items are scored from 1 (never) to 5 (always) except from items 1 and 9 (reverse). Items 1 and 2 explore the level of the child's/adolescent's physical activity, energy and fitness. Items 3 and 4 cover how much the child/adolescent experiences depressive moods and emotions and stressful feelings. Items 5 and 6 ask about the child's opportunities to structure and enjoy his/her social and leisure time and participation in social activities. Item 7 explores the quality of the interaction between child/adolescent and parent or carer and the child's/adolescent's feelings toward their parents/carers. Item 8 examines the nature of the child's/adolescent's relationships with other children/adolescents. Finally, items 9 and 10 explore the child's/adolescent's perception of his/ her cognitive capacity and satisfaction with school performance. Higher score is better
Warwick-Edinburgh Mental Well-being Scale (WEMWBS) | Baseline and 12 months
  WEMWBS is a 7 item measure of maternal mental health. A total score is calculated by summing the 7 items and converting the raw score according to a published conversion table. Score range 7- 35 for both raw and converted scores. High score is better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: maiken Pontoppidan, Principal Investigator — VIVE
Locations (3):
- Denmark (3):
  - FDF, Copenhagen
  - KFUM spejderne, Copenhagen
  - KFUMs sociale arbejde, Strib

IPD SHARING:
Plan to Share IPD: Undecided
Depending on the number of participants and the information provided we will decide if individual participant data can be made available or not

REFERENCES:
- [Derived] Pontoppidan M, Thorsager M, Larsen AT, Friis-Hansen M. Family Club Denmark: A Quasi-Randomized Study of a Volunteer-Based Intervention to Support Vulnerable Families. Healthcare (Basel). 2024 May 29;12(11):1115. doi: 10.3390/healthcare12111115. PMID 38891190
- [Derived] Pontoppidan M, Thorsager M, Larsen AT, Friis-Hansen M. Family Club Denmark #strongertogether - a volunteer intervention for disadvantaged families: study protocol for a quasi-experimental trial. BMC Psychol. 2020 Jun 1;8(1):55. doi: 10.1186/s40359-020-00426-0. PMID 32487180